CLINICAL TRIAL: NCT04571814
Title: An Investigation of a Parent/Child Psycho-social Computerized Intervention Targeting the Error-related Negativity in Young Children
Brief Title: Targeting the ERN Computerized Intervention Targeting the Error-related Negativity in Young Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Florida State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Alexandria Meyer, Assistant Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00000605; 5K01MH117366-02 (NIH)
Record Dates: First submitted 2020-09-17; First posted 2020-10-01 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Anxiety
Keywords: error-related negativity; anxiety disorders; performance anxiety; perfectionism
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Parent and child intervention (Experimental): Both parent and child will receive a computerized intervention to reduce error sensitivity.
  Interventions: Behavioral: Psycho-social, computerized intervention targeting error sensitivity
- Parent intervention and child control (Experimental): Parent will receive a computerized intervention to reduce error sensitivity and child will receive an active control (a computerized program targeting health behaviors).
  Interventions: Behavioral: Psycho-social, computerized intervention targeting error sensitivity
- Parent control and child intervention (Experimental): Child will receive a computerized intervention to reduce error sensitivity and parent will receive an active control (a computerized program targeting health behaviors).
  Interventions: Behavioral: Psycho-social, computerized intervention targeting error sensitivity
- Parent and child control (Active Comparator): Both parent and child will receive an active control (a computerized program targeting health behaviors).
  Interventions: Behavioral: Psycho-social, computerized intervention targeting error sensitivity

INTERVENTIONS:
Behavioral: Psycho-social, computerized intervention targeting error sensitivity — A psycho-social, computerized intervention for parents and children targeting error sensitivity. This intervention will be based on the constructs in the Child Error Sensitivity Index, as well as other constructs, that relate to the error-related negativity - for example, perfectionism, fear of evaluation from others, and over-valuation of the negative consequences of errors. The parent version of the intervention will include these same basic concepts, but will also target parenting style and provide psychoeducation on the negative impact of over-reacting to children's mistakes.
  The parent version will also include examples of how to model appropriate reactivity to mistakes, and provide video vignettes and examples of both critical and adaptive parenting reactions to mistakes.

SUMMARY:
Anxiety disorders are the most common form of psychopathology, frequently begin in childhood, and are often associated with substantial lifelong impairment2. Thus, there is a critical need and opportunity to identify neural markers of risk that distinguish anxious from healthy trajectories early in development that may serve as novel targets for intervention - especially if they are evident before symptoms have become impairing. One promising neural marker of anxiety is increased brain activity in response to mistakes, as reflected by the error-related negativity (ERN). Considering that the ERN is elevated before anxiety symptoms become impairing, it is critical to identify environmental factors that may shape the ERN early in life - so that those factors can be manipulated to reduce the ERN and potentially mitigate risk. In a sample of 295 six-year old children, the investigators found that both observational and self-report measures of harsh parenting style related to an increased ERN in offspring. A similar pattern of results was reported by another lab among 4 year-old children. Moreover, results suggested that the ERN mediated the relationship between harsh parenting and child anxiety disorders.

Based on these data, the investigators propose to develop a novel psychosocial intervention to be administered to both parents and children, which aims to normalize the ERN in children (i.e., reduce over-reactivity to making errors). The proposed Mentored Career Development Award (K01) is designed to extend the investigator's previous work on the ERN, parenting, and risk for anxiety in young children to test the extent to which the ERN can be modulated. Specifically, the investigators will recruit 100 parent/child dyads, high in error sensitivity, and randomize 75 to an intervention condition and 25 to an active control condition. The investigators will measure the ERN in children pre and post intervention, as well as baseline anxiety symptoms. At a six-month follow-up, the investigators will assess children's ERN, as well as anxiety symptoms, to examine to what extent intervention-related changes in the ERN relate to decreases in anxiety symptoms. Moreover, this training plan builds on the investigator's expertise on the ERN and anxiety, and integrates expertise in the design and implementation of computerized interventions, as well as advanced statistical analyses related to intervention outcomes.

DETAILED DESCRIPTION:
Anxiety disorders are the most common form of psychopathology, and are associated with substantial impairment. Longitudinal-prospective work has demonstrated anxiety disorders often begin in childhood and persist across the lifespan. Therefore, there is a critical need and opportunity to identify markers of risk that predict anxious trajectories of development. Such markers may be novel targets for intervention, that are evident before symptoms become impairing. Furthermore, identifying environmental factors that impact neural markers of risk may be useful in developing interventions. One promising biomarker of anxiety is increased brain activity in response to errors, as reflected by the error-related negativity (ERN). The ERN is a deflection in the event-related potential (ERP) occurring after an individual makes a mistake on lab-based tasks. In over 45 studies to date, the ERN has been found to be increased in anxious individuals, including children as young as age 6, and has thereby been proposed as a neural biomarker of anxiety. Critically, an increased ERN has also been shown to predict the onset of new anxiety disorders in children and adolescents, even while controlling for baseline anxiety symptoms.

Considering the ERN is elevated before anxiety symptoms become impairing, it is crucial to identify factors that may modify the ERN early in life - so as to prevent the onset of clinical anxiety. Given the ERN can be potentiated in the lab with punishment for errors, the investigators hypothesized that exposure to critical parenting styles may sensitize children to their own mistakes. Indeed, the investigators did find, in a large sample of young children (295 six-year old children), that both observational and self-report measures of critical parenting style related to an increased ERN in offspring. Moreover, results suggested the ERN mediated the relationship between critical parenting and child anxiety disorders, supporting the proposition that an increased ERN may be one mechanism by which parenting impacts child anxiety. This finding has since been replicated in even younger children (approximately 4 years old), suggesting this neural risk marker for anxiety appears to be shaped by parenting behaviors, and thus, may be a modifiable biomarker. However, no previous work has examined to what extent modifying parenting may impact the ERN.

Drawing upon this recent work, in the current proposal, the investiagotors will develop a novel psychosocial intervention to be administered to both parents and children, which aims to normalize the ERN in children (i.e., reduce over-reactivity to making errors). Given recent evidence that critical parenting and parental sensitivity to children's errors relates to an increased ERN in children, combined with pilot data suggesting that the ERN can be reduced via a psychosocial intervention, the investigators will use a brief, computerized, psychosocial intervention to directly target this well-established neurobiological risk marker in children.

The proposed Mentored Career Development Award (K01) is designed to extend previous work on the ERN, parenting, and risk for anxiety in young children to test the extent to which the ERN can be modulated. Specifically, the investigators will recruit 100 parent/child dyads, high in error sensitivity, and randomize 75 to an intervention condition and 25 to an active control condition. The investigators will measure the ERN in children pre and post intervention, as well as baseline anxiety symptoms. At a six-month follow-up, the investigators will assess children's ERN, as well as anxiety symptoms, to examine to what extent intervention-related changes in the ERN relate to decreases in anxiety symptoms. Moreover, this training plan builds on the investigator's expertise on the ERN and anxiety, and integrates expertise in the design and implementation of computerized interventions, as well as advanced statistical analyses related to intervention outcomes. AIM 1: Examine whether a neural marker of risk for anxiety (i.e., the ERN) in children is decreased during a single lab visit, via a brief, computerized intervention designed to target error sensitivity. The investigators hypothesize that children that participate in the active condition will experience a decrease in the ERN at the first assessment, compared to children in the control condition. 1a. Examine whether initial intervention-related decreases in the ERN relate to decreased anxiety symptoms at the six-month follow-up. The investigators expect that the extent to which children's ERNs are normalized during the initial intervention will relate to a lasting reduction in anxiety symptoms. AIM 2: Examine whether the ERN in children in the intervention condition display a reduction in the ERN from the initial lab assessment to the six-month follow-up assessment. The investigators expect the parenting aspect of the intervention to impact children between the assessments, therefore the investigators hypothesize that children in the active condition will experience a reduction in the ERN magnitude from the first to second lab assessment. 2a. Examine whether intervention-related decreases in the ERN between the first and second assessment relate to decreases in anxiety symptoms at the six-month follow-up. The investigators hypothesize that the extent the ERN decreases from the first to the second lab assessment to relate to decreases in anxiety symptoms in children. AIM 3: Examine whether changes in the ERN, and thus changes in child anxiety, are mediated by changes in parenting style and parental sensitivity to children's errors. This exploratory aim focuses on validating the impact parenting has on child symptoms and explores to what extent a brief, computerized intervention can modulate parent behavior and thus anxiety symptoms in children.

ELIGIBILITY:
Inclusion Criteria:

Family with a child between the ages of 5 and 7 years old Parent or child must be high in error sensitivity (as measured by a self-report measure - must be at least .5 standard deviations above the mean on the Child Error Sensitivity Index)

Exclusion Criteria:

The absence of a primary caregiver that can accompany the child to the laboratory visit Either the child or the parent does not speak English

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 222 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Initial Target Engagement: the error-related negativity (ERN, a physiological EEG measure) during the first lab visit | Baseline assessment
  The error-related negativity (ERN, a physiological EEG measure) will be measured before and after a brief, computerized intervention during the first lab visit.
Target Engagement: the error-related negativity (ERN, a physiological EEG measure) at the follow-up lab visit | Follow-up assessment (6-month follow-up)
  The error-related negativity (ERN, a physiological EEG measure) will be at the 6-month follow-up lab visit.
Child anxiety symptoms at follow-up lab visit measured by the Screen for Child Anxiety Related Emotional Disorders (SCARED). | Follow-up assessment (6-month follow-up)
  We will also examine anxiety symptoms at the six-month follow-up assessment with the Screen for Child Anxiety Related Emotional Disorders (SCARED). The SCARED contains 38 items that are rated from 0 to 2, the minimum score is 0 and the maximum score is 76. A higher score indicates more anxiety symptoms (i.e., a worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Alexandria Meyer, PhD, Principal Investigator — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-19): https://cdn.clinicaltrials.gov/large-docs/14/NCT04571814/Prot_SAP_000.pdf